CLINICAL TRIAL: NCT05108636
Title: The Effect Of Therapeutic Touch and Music Rest on Sleeping Applied to Children With Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maksude YILDIRIM (Other)
Collaborators: Inonu University (Other)
Responsible Party: Sponsor-Investigator, Maksude YILDIRIM, Research Assistant, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TDK-2020-2358
Record Dates: First submitted 2021-09-09; First posted 2021-11-05 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Liver Transplant Disorder; Sleep
Keywords: Liver; Transplant; Therapeutic touch; Music; Sleep
MeSH Terms: interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Touch (Experimental): TD process:
  * After the procedure was explained, the focus was on the child to be treated,
  * Intended to help the child's treatment and sleep,
  * The patient's energy field was scanned with the hands at a distance of 8-12 cm from the patient's skin (2 times)
  * To remove the blockages determined regarding the energy flow and to facilitate the energy flow, manual cleaning was performed (2 times),
  * Imbalances in the energy fields were tried to be treated by using mental visualization techniques such as dreaming, positive thinking and visualization, by directing the universal life energy to sick individuals with calm and rhythmic hand movements (2 times),
  * Reassessed to determine whether success has been achieved in treating imbalances in the energy field.
  Interventions: Other: Therapeutic Touch
- Music Rest (Experimental): * Parents and children will be informed about the "Music Rest" before the procedure.
  * One day before the "Music Rest" practice, the child's sleep will be evaluated with "Actigraphy". Starting the day after the first measurement, the "Music Rest" will be held for three days as a 20-minute practice period per day. In order to help the child sleep, the child will be listened to music (such as lullaby, classical music) preferred by the patient or his family.
  * Before the "Music Rest" application, the patient's room will be ventilated and a spacious and quiet environment will be provided during the application.
  * The sound level of the music played will be kept between 45-65 dB.
  * Nursing interventions will be written in more detail after the data of the research is collected.
  Interventions: Other: Music Rest

INTERVENTIONS:
Other: Therapeutic Touch — Therapeutic touch; It is a low-cost, non-contra-indications, easy-to-apply and non-invasive form of complementary therapy that can be applied anywhere and at any time (Vanaki et al., 2016). Therapeutic touch was developed by Krieger in 1975 as a nursing intervention to help and even heal the patient by balancing the patient's energy field (Marta et al., 2010). The basic assumption of therapeutic touch is that people have energy fields and these energy fields interact with the environment (Hanley, 2008). Therapeutic touch aims to harmonize, renew and heal the flow of the human energy field by removing the blockages of a person's biofield (Mueller et al., 2019). Unlike other touch-based methods such as massage therapy, therapeutic touch does not require the practitioner to physically touch the patient. Instead, the practitioner uses their hands to focus their energy and intent to help the recipient (Hanley, 2008).
  Arms: Therapeutic Touch
Other: Music Rest — The use of music in the treatment of diseases has been seen in many civilizations since ancient times. In ancient Greek and Roman communities, individuals resorted to music to get rid of their humanitarian problems, while in Ancient Egypt, music was used to give strength to patients during birth (Kor & Adar, 2016). In today's studies, it has been determined that music positively affects the physiological parameters, nutrition, hospital stay and sleep of the patients (O'Toole et al., 2017; Van Der Heijden et al., 2016). It is important that the sound level is within the appropriate limits while listening to music to the patients. The American Academy of Pediatrics recommends a sound level between 45dB- a maximum of 65dB (ACOG - AAP, 2012). The World Health Organization recommends a sound level of 35 dB during the day and 30 dB at night (Berglund et al., 2000).
  Arms: Music Rest

SUMMARY:
Today, the demand for liver transplantation is increasing day by day, since liver transplantation is considered the most effective treatment for end-stage liver disease. Patients who have undergone major surgery such as liver transplantation may experience sleep-related problems due to common complications of surgical procedures. However, in some studies, it is stated that practices such as acupuncture, exercise, mindfulness, therapeutic touch, listening to music, yoga, etc., performed by nurses, reduce the sleep-related problems of patients. In this study, the effects of therapeutic touch and music on the sleep of children with liver transplantation will be examined.

DETAILED DESCRIPTION:
Liver transplantation is considered the most effective method in the treatment of end-stage liver disease. For this reason, the number of patients waiting and receiving liver transplantation is increasing day by day. While the total number of adult and pediatric patients awaiting liver transplantation in our country in 2018 was 2142, the number of patients who received transplantation was 1587, the number of patients awaiting liver transplantation in 2019 was 2261, and the number of patients with transplantation was 1776.

Patients undergoing major surgery, frequently encountered conditions such as pain caused by surgical procedures, noise in surgical clinics, stress due to surgical procedure, they may experience sleep-related problems due to concerns arising from uncertainties about the process. Rabbits et al. reported in their study that poor sleep quality associated with postoperative pain is common in children undergoing major surgery. In some studies with children who have been transferred, it has been determined that children have complaints such as irregular breathing during sleep, excessive daytime sleepiness, daytime behavior problems and restless legs. Petersen et al. determined that fatigue was seen in the majority of children with liver transplantation and this fatigue was mostly associated with sleep/rest.

Sleep is a very important process for maintaining a healthy life and human health is significantly affected in cases of insomnia or poor sleep quality. While the catabolic process is active during wakefulness, the anabolic process is activated during sleep. Considering the anabolic process during sleep, it is of great importance for patients to have a quality sleep, especially after surgical intervention, in order to regain their old health. However, studies show that major surgical interventions cause deterioration in sleep quality. With good nursing care after the surgical procedure, patients can have a quality sleep. In some studies, it is stated that complementary and alternative treatment methods such as acupuncture, exercise, mindfulness, therapeutic touch, listening to music, yoga affect sleep positively. One of these complementary and alternative treatment methods is therapeutic touch. Therapeutic touch (TD) is based on the assumption that humans have energy fields and that these energy fields interact with the environment. In addition, therapeutic touch advocates the idea that there are imbalances in the energy fields of the sick individuals and that these imbalances can be corrected with the application of TD and contribute to the healing process. Efendi et al., in their study with preterm infants, determined that therapeutic touch and listening to the mother's voice increase the sleep quality of preterm infants. Hedlund et al., in their study with children with fontan (single ventricle) circulation, determined that exercise increased sleep quality. When the literature was examined, only one study was found to improve the sleep quality of children who had undergone surgery. In addition, no study has been found in the literature examining the effect of therapeutic touch on the sleep of children with liver transplantation. In this study, the effects of therapeutic touch and music on the sleep of children with liver transplantation will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Being within a period of at least one month and at most two years after the transplant
* 0-18 years old
* Conscious
* spontaneous breathing
* No hearing problems
* Pain free
* Children who do not use sleeping pills will be included in the study.

Exclusion Criteria:

* Children with pain
* Children using sleeping pills

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
The effect of therapeutic touch on sleep | 10 months
  The actigraphy device, which can be easily attached to the wrist of the patients, is used to evaluate and document the physical movements of the patients related to sleep. The device can keep a record of the patient's activity for 24 hours. The patient's information can be read and evaluated with the help of a special software of the device.
  After measuring the sleep of the patients with the actigraphy device for 24 hours, therapeutic touch will be applied for 3 days and at the end of the 3rd day, their sleep will be measured again with the actigraphy device for 24 hours.
The effect of music on sleep | 10 months
  The actigraphy device, which can be easily attached to the wrist of the patients, is used to evaluate and document the physical movements of the patients related to sleep. The device can keep a record of the patient's activity for 24 hours. The patient's information can be read and evaluated with the help of a special software of the device.
  After the patients' sleep is measured with an actigraphy device for 24 hours, they will listen to music they want for 3 days, and at the end of the 3rd day, their sleep will be measured again with an actigraphy device for 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Emriye Hilal YAYAN, PhD, Study Director — Inönü University; Maksude YILDIRIM, Msc, Principal Investigator — Inönü University
Locations (1):
- Inönü University, Malatya, Battalgazi, Turkey (Türkiye)

DOCUMENTS (3):
  • Study Protocol (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT05108636/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT05108636/SAP_001.pdf
  • Informed Consent Form (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT05108636/ICF_002.pdf